CLINICAL TRIAL: NCT04846153
Title: Comparing Human and Computer-based Quantification of Airway Stenosis From Bronchoscopic Images
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Nobuhiko Hata, PhD, Professor of Radiology, Brigham and Women's Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: AirwayStenosis2021
Record Dates: First submitted 2021-04-12; First posted 2021-04-15 (Actual); Last update posted 2021-04-15 (Actual); Status verified 2021-04

CONDITIONS: Airway Obstruction
Keywords: Airway Stenosis; Stenosis Index Quantification
MeSH Terms: conditions — Airway Obstruction

STUDY DESIGN:
Intervention Model Description: Physicians enrolling the study are exclusively assigned to Human-based Quantification.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Human-based Quantification (Other): No intervention. No support tool will be used for quantifying airway stenosis from the bronchoscopic images collected previously.
  Interventions: Other: Human-based Quantification of Airway Stenosis
- Computer-based Quantifiction (Active Comparator): Computer based support tool will quantifying airway stenosis from the bronchoscopic images collected previously.
  Interventions: Device: Computer-based Quantification of Airway Stenosis From Bronchoscopic Images.

INTERVENTIONS:
Other: Human-based Quantification of Airway Stenosis — Human-based Quantification of Airway Stenosis From Bronchoscopic Images.
  Arms: Human-based Quantification
Device: Computer-based Quantification of Airway Stenosis From Bronchoscopic Images. — Computer-based Quantification of Airway Stenosis From Bronchoscopic Images.
  Arms: Computer-based Quantifiction

SUMMARY:
This is a pilot study to assess the utility of the automatic stenosis index quantification using 3D Slicer software (Computer-based Quantification). We will recruit three physicians to perform a similar analysis using video images of the same bronchoscopes images (Human-based Quantification). This study relates to the latter data collection.

ELIGIBILITY:
Inclusion Criteria:

* Physicians who are trained in bronchoscopy.
* Physicians who are willing and able to understand the scope of the study.

Exclusion Criteria:

* Physicians who are not trained in bronchoscopy.
* Physicians who are unwilling and unable to understand the study procedure
* Employees under the direct supervision of the investigators conducting the research

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 3 (Estimated)
Dates: Start 2021-04-16 (Estimated); Primary Completion 2021-04-16 (Estimated); Study Completion 2021-07-16 (Estimated)

PRIMARY OUTCOMES:
Stenosis index quantified [0-100%] | 1 year
  The stenosis index quantified subjectively by the physician, defined ration between cross-sectional area of the obstructed airway and that of a normal airway.

IPD SHARING:
Plan to Share IPD: No
Currently, there is no plan to share IPD.